CLINICAL TRIAL: NCT00449644
Title: A Phase II, Placebo-controlled, Double-blind, Randomized Trial to Evaluate the Anti-bacterial Activity, Safety, and Tolerability of TMC207 in Subjects With Newly Diagnosed Sputum Smear-positive Pulmonary Infection With Multi-drug Resistant Mycobacterium Tuberculosis (MDR-TB).
Brief Title: TMC207-TiDP13-C208: Anti-bacterial Activity, Safety, and Tolerability of TMC207 in Participants With Multi-drug Resistant Mycobacterium Tuberculosis (MDR-TB).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Infectious Diseases BVBA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR011929; TMC207-TIDP13-C208 (Other: Janssen Infectious Diseases BVBA); 2007-004462-40 (EudraCT Number); NCT00614627 (obsolete NCT alias); NCT00980265 (obsolete NCT alias)
Record Dates: First submitted 2007-03-16; First posted 2007-03-20 (Estimated); Results first posted 2013-06-25 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; MDR TB
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Multidrug-Resistant | interventions — bedaquiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- TMC207 Stage 1 (Experimental): TMC207 400mg (4 tablets) once daily for 14 days, 200mg (2 tablets) three times a week for 6 weeks in addition to Background Regimen (BR) for multi-drug resistant tuberculosis (MDR-TB).
  Interventions: Drug: TMC207; Drug: Background regimen (BR) for MDR-TB (multi-drug resistant tuberculosis)
- Placebo Stage 1 (Placebo Comparator): Placebo 4 tablets once daily for 14 days, 2 tablets three times a week for 6 weeks in addition to BR for MDR-TB.
  Interventions: Drug: Placebo; Drug: Background regimen (BR) for MDR-TB (multi-drug resistant tuberculosis)
- TMC207 Stage 2 (Experimental): TMC207 400mg (4 tablets) once daily for 14 days, 200mg (2 tablets) three times a week for 22 weeks in addition to BR for MDR-TB.
  Interventions: Drug: TMC207; Drug: Background regimen (BR) for MDR-TB (multi-drug resistant tuberculosis)
- Placebo Stage 2 (Placebo Comparator): Placebo 4 tablets once daily for 14 days, 2 tablets three times a week for 22 weeks in addition to BR for MDR-TB.
  Interventions: Drug: Placebo; Drug: Background regimen (BR) for MDR-TB (multi-drug resistant tuberculosis)

INTERVENTIONS:
Drug: TMC207 — TMC207 400mg (4 tablets) once daily for 14 days, 200mg (2 tablets) three times a week for 6 or 22 weeks.
  Arms: TMC207 Stage 1; TMC207 Stage 2
Drug: Placebo — Placebo 4 tablets once daily for 14 days, 2 tablets three times a week for 6 or 22 weeks.
  Arms: Placebo Stage 1; Placebo Stage 2
Drug: Background regimen (BR) for MDR-TB (multi-drug resistant tuberculosis) — Background Regimen (BR) of antibacterial drugs used in the treatment of TB according to national TB program and selected at the baseline visit as speciified in the protocol for up to 96 weeks.

SUMMARY:
The objective of this study is to demonstrate that the antibacterial activity of TMC207 is better than placebo when added to a standardized Background Regimen (BR) for treatment of multi-drug resistant TB. Also safety and tolerability will be evaluated.

DETAILED DESCRIPTION:
The trial will be conducted in 2 consecutive stages, an exploratory (investigative) stage (Stage 1) and a proof of effectiveness stage (Stage 2). During Stage 1, a panel of 50 participants will be randomized (participants are assigned different treatments based on chance) to receive either TMC207 or placebo for 8 weeks on top of a BR. In Stage 2, another panel of 150 participants will be randomized to receive either TMC207 or placebo for 24 weeks on top of a BR. TMC207 will be dosed as 400 mg every day for the first 2 weeks, and as 200 mg 3 times/week for the following 6 or 22 weeks during Stages 1 and 2, respectively. When the participants in Stage 1 have completed 8 weeks double-blind (neither theparticipant nor the physician knows whether drug or placebo is being taken, or at what dosage) treatment with TMC207 or placebo (or have discontinued earlier), the primary Stage 1 analysis will be performed on all data of the first 8 weeks of treatment. Following this Stage 1 analysis, Stage 2 will be initiated and a panel of 150 new participants will be enrolled. After the double-blind treatment phase in both Stage 1 and Stage 2, participants will continue to receive MDR-TB treatment as per national treatment guidelines. They will be followed for safety, tolerability, pharmacokinetics, and microbiological efficacy for 96 weeks after receiving their last dose of TMC207 or placebo. The Data Safety Monitoring Board Committee will review these data on a regular basis. The DSMB/DSMC is a group of experts in tuberculosis and clinical trial conduct who have no commercial interests in the development of TMC207 and the company (Tibotec, BVBA) that is developing the new TB drug.

ELIGIBILITY:
Inclusion Criteria:

* Females of non-childbearing potential
* Patients with newly diagnosed sputum smear-positive pulmonary MDR-TB infection
* Patients must consent to HIV-testing
* Patients must be willing to discontinue all TB drugs to allow 7 days washout
* Patients having normal weight
* Patients are willing to be hospitalized per standard of care.

Exclusion Criteria:

* Previously having been treated for MDR-TB
* Having a significant cardiac arrhythmia that requires medication
* For HIV infected patients, having a CD4+ count < 300 cells/µL
* Patients with complicated or severe extrapulmonary manifestations of TB or neurological manifestations of TB
* Patients who will require surgical procedure for management of their TB
* Evidence of chorioretinitis, optic neuritis, or uveitis at screening
* Having had a drug susceptibility test performed prior to screening and being not susceptible to at least 3 of the 5 classes of TB drugs used to treat MDR-TB
* Women who are pregnant and/or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2007-06; Primary Completion 2010-03 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Infectious Diseases BVBA Clinical Trial, Study Director — Janssen Infectious Diseases BVBA
Locations (16):
- Rio de Janeiro, Brazil
- India (2):
  - Chennai
  - New Delhi
- Stopinu Region, Latvia
- Lima, Peru
- Quezon City, Philippines
- Moscow, Russia
- South Africa (6):
  - Bethelsdorp
  - Cape Town
  - Durban
  - George
  - Klerksdorp
  - Sandringham
- Thailand (3):
  - Chiang Mai
  - Nakhon
  - Nonthaburi

REFERENCES:
- [Result] Diacon AH, Pym A, Grobusch M, Patientia R, Rustomjee R, Page-Shipp L, Pistorius C, Krause R, Bogoshi M, Churchyard G, Venter A, Allen J, Palomino JC, De Marez T, van Heeswijk RP, Lounis N, Meyvisch P, Verbeeck J, Parys W, de Beule K, Andries K, Mc Neeley DF. The diarylquinoline TMC207 for multidrug-resistant tuberculosis. N Engl J Med. 2009 Jun 4;360(23):2397-405. doi: 10.1056/NEJMoa0808427. PMID 19494215
- [Derived] Bolhuis MS, Akkerman OW, Sturkenboom MGG, van Boven JFM, Alffenaar JC, Stevens J. Bedaquiline exposure in people with drug-resistant TB treated for diabetes: analysis of two phase 2 trials. Int J Tuberc Lung Dis. 2023 Apr 1;27(4):335-337. doi: 10.5588/ijtld.22.0581. No abstract available. PMID 37035978
- [Derived] Meyvisch P, Kambili C, Andries K, Lounis N, Theeuwes M, Dannemann B, Vandebosch A, Van der Elst W, Molenberghs G, Alonso A. Evaluation of six months sputum culture conversion as a surrogate endpoint in a multidrug resistant-tuberculosis trial. PLoS One. 2018 Jul 19;13(7):e0200539. doi: 10.1371/journal.pone.0200539. eCollection 2018. PMID 30024924
- [Derived] Pym AS, Diacon AH, Tang SJ, Conradie F, Danilovits M, Chuchottaworn C, Vasilyeva I, Andries K, Bakare N, De Marez T, Haxaire-Theeuwes M, Lounis N, Meyvisch P, Van Baelen B, van Heeswijk RP, Dannemann B; TMC207-C209 Study Group. Bedaquiline in the treatment of multidrug- and extensively drug-resistant tuberculosis. Eur Respir J. 2016 Feb;47(2):564-74. doi: 10.1183/13993003.00724-2015. Epub 2015 Dec 2. PMID 26647431
- [Derived] Diacon AH, Pym A, Grobusch MP, de los Rios JM, Gotuzzo E, Vasilyeva I, Leimane V, Andries K, Bakare N, De Marez T, Haxaire-Theeuwes M, Lounis N, Meyvisch P, De Paepe E, van Heeswijk RP, Dannemann B; TMC207-C208 Study Group. Multidrug-resistant tuberculosis and culture conversion with bedaquiline. N Engl J Med. 2014 Aug 21;371(8):723-32. doi: 10.1056/NEJMoa1313865. PMID 25140958

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial consisted of an exploratory stage (Stage 1) and a proof-of-efficacy stage (Stage 2). Different participants were enrolled in each stage. Participants in Stage 2 who met protocol-specified criteria were offered open-label treatment with TMC207 after Week 24 (ie, rollover arm).
Pre-assignment Details: A total of 208 participants were randomized and 207 (47 participants in Stage 1 and 160 participants in Stage 2) started treatment with placebo or TMC207 (1 participant did not receive study drug). One placebo participant in Stage 2 rolled-over to treatment with TMC207 after Week 24.
Groups:
- TMC207 / BR (Stage 1): Weeks 1 and 2: 400 mg TMC207 once daily administered as 4 tablets, and Background Regimen (BR) for Multi-drug resistant tuberculosis (MDR-TB). Week 3 to 8: 200 mg TMC207 three times per week administered as 2 tablets, and BR. Only BR after Week 8.
- Placebo / BR (Stage 1): Weeks 1 and 2: Placebo once daily administered as 4 tablets, and Background Regimen (BR) for Multi-drug resistant tuberculosis (MDR-TB). Week 3 to 8: Placebo three times per week administered as 2 tablets, and BR. Only BR after Week 8.
- TMC207 / BR (Stage 2): Weeks 1 and 2: 400 mg TMC207 once daily administered as 4 tablets, and Background Regimen (BR) for Multi-drug resistant tuberculosis (MDR-TB). Week 3 to 24: 200 mg TMC207 three times per week administered as 2 tablets, and BR. Only BR after Week 24.
- Placebo / BR (Stage 2): Weeks 1 and 2: Placebo once daily administered as 4 tablets, and Background Regimen (BR) for Multi-drug resistant tuberculosis (MDR-TB). Week 3 to 24: Placebo three times per week administered as 2 tablets, and BR. Only BR after Week 24.
Period: Overall Study
Arm/Group | TMC207 / BR (Stage 1) | Placebo / BR (Stage 1) | TMC207 / BR (Stage 2) | Placebo / BR (Stage 2)
Started | 23 | 24 | 79 | 81
Rollover | 0 | 0 | 0 | 1
Completed | 13 | 11 | 50 | 49 (After Week 24, 1 patient rolled over to treatment with TMC207 and was not completed or discontinued.)
Not Completed | 10 | 13 | 29 | 32
Not completed — Adverse Event | 0 | 0 | 3 | 5
Not completed — Death | 1 | 0 | 6 | 1
Not completed — Lost to Follow-up | 1 | 1 | 5 | 3
Not completed — Pregnancy | 0 | 0 | 3 | 2
Not completed — Protocol Violation | 4 | 4 | 3 | 7
Not completed — Withdrawal by Subject | 3 | 4 | 6 | 7
Not completed — Inclusion/exclusion criteria not met | 0 | 0 | 2 | 6
Not completed — Other | 1 | 4 | 1 | 0
Not completed — Rolled-over to treatment with TMC207 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TMC207 / BR (Stage 1) | Placebo / BR (Stage 1) | TMC207 / BR (Stage 2) | Placebo / BR (Stage 2) | Total
Number analyzed (Participants) | 23 | 24 | 79 | 81 | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (11.66) | 33.6 (11.04) | 36.2 (13.13) | 35.8 (11.01) | 35.7 (11.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 27 | 32 | 71
  Male | 18 | 17 | 52 | 49 | 136

OUTCOME MEASURES:

1. Primary Outcome: The Time to Sputum Culture Conversion at Week 8 (Stage 1)
Description: The table below shows the time to sputum culture conversion. Sputum culture conversion is defined as as having 2 consecutive negative cultures at least 25 days apart, not followed by a confirmed positive during the considered time period. Participants who discontinue or die during the considered time period are considered as non-responders and censored at their last assessment.
Time Frame: Week 8, Stage 1
Population: The modified intent-to-treat (mITT) population used for all efficacy analyses included all randomized participants who received at least 1 dose of study drug and did not have extensively drug resistant tuberculosis (XDR-TB) or non-multi-drug resistant tuberculosis (non-MDR-TB) at the start of the trial and were evaluable for efficacy.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- TMC207 / BR (Stage 1): Weeks 1 and 2: 400 mg TMC207 once daily administered as 4 tablets, and Background Regimen (BR) for Multi-drug resistant tuberculosis (MDR-TB). Week 3 to 8: 200 mg TMC207 three times a week administered as 2 tablets, and BR. Only BR after Week 8.
Arm/Group | TMC207 / BR (Stage 1) | Placebo / BR (Stage 1)
Number analyzed (Participants) | 21 | 23
Days | 51 [30 to NA] — The curve of the upper limit around the time to response curve does not cross 50%. | NA [NA to NA] — The Kaplan-Meier curve of time to response does not cross the 50% line for Placebo.
Statistical Analysis 1: Comparison: TMC207 / BR (Stage 1) vs Placebo / BR (Stage 1); Test type: Superiority or Other; p = 0.0034, Cox proportional hazards model; Treatment, lung cavitation and pooled center were used as covaritates; Hazard Ratio (HR) = 11.77, 95% CI 2-sided [2.26 to 61.23]

2. Primary Outcome: The Time to Sputum Culture Conversion at Week 24 (Stage 2)
Description: as for outcome 1
Time Frame: Week 24, Stage 2
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Placebo / BR (Stage 2): Weeks 1 and 2: Placebo once daily administered as 4 tablets, and Background Regimen (BR) for Multi-drug resistant tuberculosis (MDR-TB). Week 3 to 24: 200 mg TMC207 three times per week administered as 2 tablets, and BR. Only BR after Week 24.
Arm/Group | TMC207 / BR (Stage 2) | Placebo / BR (Stage 2)
Number analyzed (Participants) | 66 | 66
Days | 83 [56 to 97] | 125 [98 to 168]
Statistical Analysis 1: Comparison: TMC207 / BR (Stage 2) vs Placebo / BR (Stage 2); Test type: Superiority or Other; p < 0.0001, Cox proportional hazards model; Treatment, lung cavitation and pooled center were used as covaritates; Hazard Ratio (HR) = 2.44, 95% CI 2-sided [1.57 to 3.80]

3. Secondary Outcome: The Time to Sputum Culture Conversion at Week 24 (Stage 1)
Description: as for outcome 1
Time Frame: Week 24, Stage 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | TMC207 / BR (Stage 1) | Placebo / BR (Stage 1)
Number analyzed (Participants) | 21 | 23
Days | 70 [49 to 100] | 126 [98 to 134]
Statistical Analysis 1: Comparison: TMC207 / BR (Stage 1) vs Placebo / BR (Stage 1); Test type: Superiority or Other; p = 0.0022, Cox-proportional hazards model; Treatment, lung cavitation and pooled center were used as covaritates; Odds Ratio (OR) = 3.14, 95% CI 2-sided [1.51 to 6.53]

4. Secondary Outcome: The Time to Sputum Culture Conversion at Week 72 (Stage 2)
Description: as for outcome 1
Time Frame: Week 72, Stage 2
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | TMC207 / BR (Stage 2) | Placebo / BR (Stage 2)
Number analyzed (Participants) | 66 | 66
Days | 86 [70 to 99] | 168 [112 to 345]
Statistical Analysis 1: Comparison: TMC207 / BR (Stage 2) vs Placebo / BR (Stage 2); MGIT negative (Responders); Test type: Superiority or Other; p = 0.0290, Cox proportional hazards model; Treatment, lung cavitation and pooled center were used as covaritates; Odds Ratio (OR) = 1.65, 95% CI 2-sided [1.05 to 2.59]

5. Secondary Outcome: The Percentage of Participants With Sputum Culture Conversion (Stage 1)
Description: The table below shows the percentage of participants in Stage 1 who were responders to treatment. Sputum culture conversion is defined as as having 2 consecutive negative cultures at least 25 days apart, not followed by a confirmed positive during the considered time period. Participants who discontinue or die during the considered time period are considered as non-responders.
Time Frame: Week 8, 24, and 104 (Stage 1)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Groups:
- Placebo / BR (Stage 1): Weeks 1 and 2: Placebo once daily administered as 4 tablets, and Background Regimen (BR) for Multi-drug resistant tuberculosis (MDR-TB). Week 3 to 8: Placebo three times per week administered as 2 tablets, and BR. Only BR after Week.
Arm/Group | TMC207 / BR (Stage 1) | Placebo / BR (Stage 1)
Number analyzed (Participants) | 21 | 23
Percentage of Participants
  Week 8 | 47.6 | 8.7
  Week 24 | 81.0 | 65.2
  Week 104 (Stage 1 Trial End) | 52.4 | 43.5
Statistical Analysis 1: Comparison: TMC207 / BR (Stage 1) vs Placebo / BR (Stage 1); Week 8; Test type: Superiority or Other; p = 0.003, Regression, Logistic; Treatment as covariate; Risk Difference (RD) = 38.9, 95% CI 2-sided [13.97 to 63.88], Standard Error of Mean 12.38
Statistical Analysis 2: Comparison: TMC207 / BR (Stage 1) vs Placebo / BR (Stage 1); Week 24; Test type: Superiority or Other; p = 0.237, Regression, Logistic; Treatment as covariate; Risk Difference (RD) = 15.7, 95% CI 2-sided [-10.70 to 42.17], Standard Error of Mean 13.12
Statistical Analysis 3: Comparison: TMC207 / BR (Stage 1) vs Placebo / BR (Stage 1); Week 104 (Stage 1 Trial End); Test type: Superiority or Other; p = 0.5564, Regression, Logistic; Treatment as covariate; Risk Difference (RD) = 8.9, 95% CI 2-sided [-21.37 to 39.18], Standard Error of Mean 15.02

6. Secondary Outcome: The Percentage of Participants With Sputum Culture Conversion (Stage 2)
Description: The table below shows the percentage of participants in Stage 2 who were responders to treatment. Sputum culture conversion is defined as as having 2 consecutive negative cultures at least 25 days apart, not followed by a confirmed positive during the considered time period. Participants who discontinue or die during the considered time period are considered as non-responders.
Time Frame: Week 24, Week 72, and Week 120 (Stage 2)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Groups:
- TMC207 / BR (Stage 2): Weeks 1 and 2: 400 mg TMC207 once daily administered as 4 tablets, and Background Regimen (BR) for Multi-drug resistant tuberculosis (MDR-TB). Week 3 to 8: 200 mg TMC207 three times a week administered as 2 tablets, and BR. Only BR after Week 8.
- Placebo / BR (Stage 2): Weeks 1 and 2: Placebo once daily administered as 4 tablets, and Background Regimen (BR) for Multi-drug resistant tuberculosis (MDR-TB). Week 3 to 8: Placebo three times per week administered as 2 tablets, and BR. Only BR after Week 8.
Arm/Group | TMC207 / BR (Stage 2) | Placebo / BR (Stage 2)
Number analyzed (Participants) | 66 | 66
Percentage of Participants
  Week 24 | 78.8 | 57.6
  Week 72 | 71.2 | 56.1
  Week 120 | 62.1 | 43.9
Statistical Analysis 1: Comparison: TMC207 / BR (Stage 2) vs Placebo / BR (Stage 2); Week 24; Test type: Superiority or Other; p = 0.008, Regression, Logistic; Treatment as covariate; Risk Difference (RD) = 21.2, 95% CI 2-sided [5.59 to 36.83], Standard Error of Mean 7.90
Statistical Analysis 2: Comparison: TMC207 / BR (Stage 2) vs Placebo / BR (Stage 2); Week 72; Test type: Superiority or Other; p = 0.069, Regression, Logistic; Treatment as covariate; Risk Difference (RD) = 15.2, 95% CI 2-sided [-1.21 to 31.51], Standard Error of Mean 8.27
Statistical Analysis 3: Comparison: TMC207 / BR (Stage 2) vs Placebo / BR (Stage 2); Week 120; Test type: Superiority or Other; p = 0.035, Regression, Logistic; Treatment as covariate; Risk Difference (RD) = 18.2, 95% CI 2-sided [1.28 to 35.08], Standard Error of Mean 8.54

ADVERSE EVENTS:
Time Frame: Stage 1: Adverse Events were collected from 05-Jun-2007 to 04-Dec-2009. Stage 2: Adverse events were collected from 23-Apr-2008 to 31-Jan-2012.
Description: Treatment-Emergent Adverse Events (TEAE) from overall treatment phase are reported. Only patients who had at least one of the TEAEs are listed in the Other (non Serious) Adverse Event table are included in the total number of patients with Non-Serious Adverse Events.
Arm/Group | TMC207 / BR (Stage 1) | Placebo / BR (Stage 1) | TMC207 / BR (Stage 2) | Placebo / BR (Stage 2)
Serious Adverse Events (participants affected / at risk) | 1/23 | 1/24 | 18/79 | 15/81
Other Adverse Events (participants affected / at risk) | 21/23 | 23/24 | 75/79 | 75/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TMC207 / BR (Stage 1) (N=23) | Placebo / BR (Stage 1) (N=24) | TMC207 / BR (Stage 2) (N=79) | Placebo / BR (Stage 2) (N=81)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Conductive deafness (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Bronchiectasis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 2 | 1
Pyothorax (Infections and infestations) | 0 | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 2 | 3
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Surgery (Surgical and medical procedures) | 0 | 0 | 0 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TMC207 / BR (Stage 1) (N=23) | Placebo / BR (Stage 1) (N=24) | TMC207 / BR (Stage 2) (N=79) | Placebo / BR (Stage 2) (N=81)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 6 | 3
Deafness (Ear and labyrinth disorders) | 1 | 1 | 5 | 4
Deafness bilateral (Ear and labyrinth disorders) | 3 | 3 | 5 | 7
Deafness unilateral (Ear and labyrinth disorders) | 3 | 5 | 10 | 7
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 4 | 3
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 3 | 11
Visual acuity reduced (Eye disorders) | 0 | 0 | 5 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 6 | 6
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 10 | 8
Constipation (Gastrointestinal disorders) | 1 | 1 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 5 | 15
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 4 | 12
Gastritis (Gastrointestinal disorders) | 0 | 0 | 9 | 16
Nausea (Gastrointestinal disorders) | 6 | 1 | 32 | 30
Vomiting (Gastrointestinal disorders) | 1 | 3 | 23 | 22
Chest pain (General disorders) | 0 | 2 | 10 | 8
Fatigue (General disorders) | 0 | 0 | 6 | 1
Injection site pain (General disorders) | 0 | 0 | 9 | 10
Non-cardiac chest pain (General disorders) | 2 | 2 | 2 | 0
Pain (General disorders) | 0 | 0 | 2 | 6
Pyrexia (General disorders) | 0 | 1 | 8 | 7
Influenza (Infections and infestations) | 1 | 0 | 6 | 9
Nasopharyngitis (Infections and infestations) | 0 | 1 | 11 | 4
Pharyngitis (Infections and infestations) | 0 | 1 | 6 | 5
Urinary tract infection (Infections and infestations) | 0 | 0 | 5 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 4 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 5 | 2
Blood uric acid increased (Investigations) | 1 | 2 | 5 | 3
Transaminases increased (Investigations) | 0 | 0 | 5 | 0
Weight decreased (Investigations) | 0 | 0 | 3 | 5
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 9 | 6
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 3 | 20 | 27
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 29 | 22
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 9 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 6 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4 | 2 | 3
Dizziness (Nervous system disorders) | 3 | 2 | 11 | 11
Headache (Nervous system disorders) | 2 | 2 | 23 | 18
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 4 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 4 | 4
Depression (Psychiatric disorders) | 0 | 0 | 3 | 7
Insomnia (Psychiatric disorders) | 0 | 1 | 13 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 7 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 15 | 13
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 4
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 11 | 15
Rash (Skin and subcutaneous tissue disorders) | 2 | 4 | 6 | 4

LIMITATIONS AND CAVEATS:
In Participant Flow, deaths occurring during the trial are reported. In addition, 1 TMC207 and 2 placebo subjects in stage 1 and 4 TMC207 and 1 placebo subject in stage 2 died after discontinuation during long-term survival follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
It is the policy of the sponsor not to allow the investigators to publish their results or findings prior to the sponsor's publication of the overall trial results.The investigator agrees that before he/she publishes any results of this trial, he/she shall provide the sponsor with at least 45 days for full review of the prepublication manuscript prior to submission of the manuscript to the publisher.